CLINICAL TRIAL: NCT01643499
Title: A Genotype-guided Dosing Study of mFOLFIRINOX in Previously Untreated Patients With Advanced Gastrointestinal Malignancies
Brief Title: Genotype-guided Dosing of mFOLFIRINOX Chemotherapy in Patients With Previously Untreated Advanced Gastrointestinal Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0033; NCI-2012-00585 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Adenocarcinoma of the Gallbladder; Adenocarcinoma of Unknown Primary; Adult Primary Cholangiocellular Carcinoma; Advanced Adult Primary Liver Cancer; Cholangiocarcinoma of the Extrahepatic Bile Duct; Cholangiocarcinoma of the Gallbladder; Diffuse Adenocarcinoma of the Stomach; Duct Cell Adenocarcinoma of the Pancreas; Intestinal Adenocarcinoma of the Stomach; Localized Unresectable Adult Primary Liver Cancer; Metastatic Carcinoma of Unknown Primary; Metastatic Extrahepatic Bile Duct Cancer; Mixed Adenocarcinoma of the Stomach; Mucinous Adenocarcinoma of the Colon; Mucinous Adenocarcinoma of the Rectum; Newly Diagnosed Carcinoma of Unknown Primary; Signet Ring Adenocarcinoma of the Colon; Signet Ring Adenocarcinoma of the Rectum; Stage III Pancreatic Cancer; Stage IIIA Colon Cancer; Stage IIIA Gallbladder Cancer; Stage IIIA Gastric Cancer; Stage IIIA Rectal Cancer; Stage IIIB Colon Cancer; Stage IIIB Gallbladder Cancer; Stage IIIB Gastric Cancer; Stage IIIB Rectal Cancer; Stage IIIC Colon Cancer; Stage IIIC Gastric Cancer; Stage IIIC Rectal Cancer; Stage IV Gastric Cancer; Stage IV Pancreatic Cancer; Stage IVA Colon Cancer; Stage IVA Gallbladder Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Gallbladder Cancer; Stage IVB Rectal Cancer; Unresectable Extrahepatic Bile Duct Cancer
MeSH Terms: conditions — Neoplasms, Unknown Primary; Bile Duct Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Rectal Neoplasms | interventions — Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (mFOLFIRINOX) (Experimental): Patients receive oxaliplatin IV over 2 hours on, irinotecan hydrochloride IV over 1.5 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV continuously over 46 hours on days 1 and 15. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: oxaliplatin; Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: fluorouracil; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This study is being done to determine the dose of a chemotherapy drug (irinotecan [irinotecan hydrochloride]) that can be tolerated as part of a combination of drugs. There is a combination of chemotherapy drugs often used to treat gastrointestinal cancer, which consists of 5-FU (fluorouracil), leucovorin (leucovorin calcium), irinotecan and oxaliplatin and is known as "FOLFIRINOX". FOLFIRINOX is a current drug therapy combination (or regimen) used for people with advanced pancreatic cancer, although this combination is not Food and Drug Administration (FDA) approved for this indication. FOLFIRINOX was recently shown in a separate clinical trial to increase survival compared to another commonly used drug in pancreatic cancer called gemcitabine. FOLFIRINOX is also a reasonable regimen for those with other advanced cancers of the gastrointestinal tract, including colon cancer, rectal cancer, esophagus cancer, stomach cancer, gall bladder cancer, bile duct cancer, ampullary cancer, and cancers with an unknown primary location. The best dose of irinotecan to use in FOLFIRINOX is not known. This study will analyze one gene (uridine 5'-diphospho [UDP] glucuronosyltransferase 1 family, polypeptide A1 [UGT1A1] gene) of subjects for the presence of an alteration in that gene, which may affect how the body handles irinotecan. Genes help determine some of the investigators individual characteristics, such as eye color, height and skin tone. Genes may also determine why people get certain diseases and how medicines may affect them. The result of the genetic analysis will divide subjects into one of three groups: A, B, or C. Group A (approximately 45% of subjects) will receive the standard dose of irinotecan. Group B (approximately 45% of subjects) will receive a lower dose of irinotecan. Group C (approximately 10% of subjects) will receive an even lower dose of irinotecan

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose-limiting toxicity (DLT) rate in cycle #1 in each of two UGT1A1 genotype groups (*1*1, *1*28) using genotype-guided dosing of irinotecan as part of the modified (m) FOLFIRINOX regimen.

SECONDARY OBJECTIVES:

I. To determine the cumulative dose intensity of irinotecan achieved in each genotype group.

II. To determine the response rates by Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1) for each different disease (pancreatic cancer, biliary cancers, gastric cancer, colorectal cancer, adenocarcinoma of unknown primary) treated in the study.

OUTLINE:

Patients receive oxaliplatin intravenously (IV) over 2 hours, irinotecan hydrochloride IV over 1.5 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV continuously over 46 hours on days 1 and 15. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic pancreatic adenocarcinoma, colorectal adenocarcinoma, gastric adenocarcinoma, cholangiocarcinoma, gall bladder adenocarcinoma, ampullary carcinoma, adenocarcinoma of unclear primary (with a gastrointestinal primary suspected), or other primary gastrointestinal malignancy for which the treating physician feels that mFOLFIRINOX is a reasonable therapeutic option.
* Amendment (January 2014): only subjects with the following histologies will be eligible

Cohort # 1 (pancreatic cohort): locally advanced or metastatic pancreatic adenocarcinoma (19 subjects evaluable for the primary endpoint after the amendment)

Cohort #2 (biliary tract cohort): locally advanced or metastatic cholangiocarcinoma, gall bladder adenocarcinoma, or ampullary carcinoma (19 subjects evaluable for the primary endpoint after the amendment). Patients with adenocarcinoma of unclear primary that are most likely of biliary tract origin (in the opinion of the treating physician) will also be allowed on this cohort.

* Patients with a history of obstructive jaundice due to the primary tumor must have a metal biliary stent in place,
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1,
* Life expectancy > 3 months,
* Absolute neutrophil count (ANC) >= l500/ul,
* Hemoglobin >= 9g/dL,
* Platelets >= 100,000/ ul,
* Total bilirubin < 1.5 x upper limit of normal,
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvate transaminase (SGPT) < 2.5 x upper limit of normal for patients without liver metastases OR SGOT and SGPT < 5 x upper limit of normal for patients with liver metastases,
* Creatinine =< 1.5 x upper limit of normal,
* Measurable or non-measurable disease will be allowed,
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, up until 30 days after final study treatment; should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately,
* Patients taking substrates, inhibitors, or inducers of Cytochrome P450 3A4 (CYP3A4) should be encouraged to switch to alternative drugs whenever possible, given the potential for drug-drug interactions with irinotecan
* Signed informed consent.

Exclusion Criteria:

* Prior chemotherapy or radiation therapy for any cancer,
* Inflammatory bowel disease (Crohn's disease, ulcerative colitis),
* Diarrhea, grade 1 or greater by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, v. 4.0); pancreatic cancer patients with clinical evidence of pancreatic insufficiency must be taking pancreatic enzyme replacement,
* Neuropathy, grade 2 or greater by NCI-CTCAE, v. 4.0,
* Documented brain metastases,
* Serious underlying medical or psychiatric illnesses that would, in the opinion of the treating physician, substantially increase the risk for complications related to treatment,
* Active uncontrolled bleeding,
* Pregnancy or breastfeeding,
* Major surgery within 4 weeks,
* Previous or concurrent malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or any other cancer for which the patient has been previously treated and the lifetime recurrence risk is less than 30%,
* Patients with any polymorphism in UGT1A1 other than *1 or *28.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-03-26 (Actual); Primary Completion 2016-08-28 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
DLT rate in course 1 for each of the two most common genotype groups (*1*1 and *1*28) | 4 weeks
  To show that the DLT rate is less than 33% with at least 70-80% confidence, which is comparable to the standard 3+3 phase I design with 0 out of 3 or 1 out of 6 patients experiencing a DLT.

SECONDARY OUTCOMES:
Response rates (by RECIST 1.1) for patients with each different type of gastrointestinal malignancy | Up to 1 year
Cumulative dose intensity of irinotecan hydrochloride | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kindler, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Evanston CCOP-NorthShore University HealthSystem, Evanston, Illinois